CLINICAL TRIAL: NCT05170997
Title: Strategies to Improve Iodine Status in Early Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other); Public Health Agency (Northern Ireland) (Unknown); Dairy Council for Northern Ireland (Other)
Responsible Party: Principal Investigator, Jayne Woodside, PhD, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B20/32; EAT/5578/19 (Other Grant/Funding Number: Public Health Agency R&D fellowship)
Record Dates: First submitted 2021-11-25; First posted 2021-12-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Iodine Deficiency; Pregnancy Related
Keywords: Iodine; Pregnancy; Diet
MeSH Terms: interventions — Milk

STUDY DESIGN:
Intervention Model Description: There will be four parallel groups in this study, stratified by iodine supplementation and then randomised to milk or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Iodine Control (Active Comparator): Participants taking an iodine-containing multivitamin or supplement and randomly allocated not to receive milk supply.
  Interventions: Other: British Dietetic Association Iodine Fact Sheet.
- No Iodine Control (Active Comparator): Participants not taking an iodine-containing multivitamin or supplement and randomly allocated not to receive milk supply.
  Interventions: Other: British Dietetic Association Iodine Fact Sheet.
- Iodine Intervention (Experimental): Participants taking an iodine-containing multivitamin or supplement and randomly allocated to receive milk supply.
  Interventions: Dietary Supplement: Cows' milk; Other: British Dietetic Association Iodine Fact Sheet.
- No Iodine Intervention (Experimental): Participants not taking an iodine-containing multivitamin or supplement and randomly allocated to receive milk supply.
  Interventions: Dietary Supplement: Cows' milk; Other: British Dietetic Association Iodine Fact Sheet.

INTERVENTIONS:
Dietary Supplement: Cows' milk — Intervention groups will receive a free 12 week supply of cows' milk equating to a pint a day for study participants. Milk is provided by Lakeland dairies.
  Arms: Iodine Intervention; No Iodine Intervention
Other: British Dietetic Association Iodine Fact Sheet. — All participants will receive the British Dietetic Association Iodine fact sheet which discusses the importance of iodine and the dietary sources.

SUMMARY:
This study aims to investigate the benefit of increased intake of cows' milk during pregnancy on iodine status.

DETAILED DESCRIPTION:
Women of child bearing age, and those who are currently pregnant, have been found to be iodine deficient in the United Kingdom (UK). Dairy products are an essential source of iodine in the UK as iodised salt is not widely available. This study will ask women in the intervention group to drink approximately one pint of milk a day for 12 weeks during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* women at 6-16 weeks pregnant
* women receiving antenatal care within Belfast Health and Social Care Trust

Exclusion Criteria:

* women with known thyroid disease currently taking thyroid medication
* women with type one diabetes
* women under 18 years of age
* those unable to provide informed consent
* women with abnormal thyroid function tests at booking appointment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Urinary iodine concentration | 18 months
  Proportion of the maternal cohort who achieve WHO urinary iodine concentration(UIC) of >=150 micrograms/litre on early morning spot urinary sampling at 12 weeks post intervention.

SECONDARY OUTCOMES:
Iodine knowledge | 24 months
  Knowledge regarding iodine intake in the diet in pregnancy and into postpartum assessed using an iodine knowledge questionnaire that will be completed by participants at the beginning and the end of the study period.
Iodine intake | 24 months
  Intake of iodine rich foods at 29 weeks and postpartum in those who breastfeed will be assessed using four day food diaries at the beginning and end of the study, and validated iodine-specific food frequency questionnaires at the beginning of the study, at the end of the intervention period, six weeks after the end of the intervention period and at the end of the study.
Offspring | 24 months.
  Proportion of offspring with adequate UIC at 6-12 weeks old.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Mullan, MD, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Royal Jubilee Maternity Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT05170997/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT05170997/ICF_001.pdf